CLINICAL TRIAL: NCT02584452
Title: Randomized Controlled Trial Evaluating Postoperative Analgesia and Muscle Strength Between Single Versus Continuous Adductor Canal Block for Ambulatory ACL Reconstruction.
Brief Title: Trial Evaluating Postop Pain and Muscle Strength Among Regional Anesthesia Techniques for Ambulatory ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sobey, Assistant Professor of Anesthesiology & Pain Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151095
Record Dates: First submitted 2015-10-14; First posted 2015-10-22 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Rupture of Anterior Cruciate Ligament; Tear of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Mepivacaine; Saline Solution; Bupivacaine; Ropivacaine; Dexamethasone; Propofol; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Adductor Canal Nerve Catheter (Active Comparator): Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal continuous nerve catheter using normal saline bolus followed by 1/8% bupivacaine infusion through catheter at 8cc/h.
  Interventions: Drug: Mepivacaine; Procedure: adductor canal continuous nerve catheter; Drug: Normal Saline as bolus followed by bupivacaine; Drug: Propofol; Drug: Fentanyl
- Long Acting Single Bolus Adductor Canal Nerve Block (Active Comparator): Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine and 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve.
  Interventions: Drug: Mepivacaine; Procedure: adductor canal nerve block; Drug: ropivacaine and dexamethasone; Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Mepivacaine — 20cc of 2% mepivacaine <20 minutes prior to in room time.
  Other Names: Carbocaine, Polocaine
Procedure: adductor canal continuous nerve catheter — Placement of ultrasound guided adductor canal continuous nerve catheter
  Arms: Continuous Adductor Canal Nerve Catheter
Drug: Normal Saline as bolus followed by bupivacaine — normal saline as bolus for placement, followed by initiation of 1/8% bupivacaine infusion through adductor canal catheter at 8cc/h
  Other Names: Marcaine
  Arms: Continuous Adductor Canal Nerve Catheter
Procedure: adductor canal nerve block — ultrasound guided adductor canal nerve block
  Arms: Long Acting Single Bolus Adductor Canal Nerve Block
Drug: ropivacaine and dexamethasone — 10cc of 0.5% ropivacaine + 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve
  Other Names: Naeopin
  Arms: Long Acting Single Bolus Adductor Canal Nerve Block
Drug: Propofol — Anesthesia induction will include a propofol bolus.
  Other Names: Diprivan; Propoven
Drug: Fentanyl — Intraoperative opioid should be limited to no more than 150mcg of fentanyl.
  Other Names: Sublimaze

SUMMARY:
Despite the apparent multifaceted benefit in differentiating blockade sites and duration of nerve blockade, the efficacy of continuous adductor canal blockade utilized specifically in ACL reconstruction has not been extensively studied. This study will test the hypothesis that the use of the adductor canal continuous nerve catheter will result in lower subjective pain scores on postoperative day 2 and improved quadriceps strength on postoperative day 1.

DETAILED DESCRIPTION:
Study participants will be randomized to 2 groups: (1) continuous adductor canal nerve catheter or (2) long-acting single bolus adductor canal nerve block.

Following random selection via random envelope selection patients will receive the following procedures. Both groups will receive ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time.

Intraoperative care will consist of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert, Group 1 patients 1 will receive ultrasound guided adductor canal continuous nerve catheter using normal saline as bolus for placement, followed by initiation of 1/8% bupivacaine infusion through catheter at 8cc/h. Group 2 will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine + 2mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve14. After adequate instruction including catheter education (if applicable) patients are to be discharged home.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 and older
* Patients who are scheduled to undergo an ACL reconstruction with patella or allograft
* Patient does not have a contraindication to receiving regional anesthesia

Exclusion Criteria:

* Allergy to local anesthetics, dexamethasone, or adhesive tape
* Patients undergoing hamstring graft for ACL
* Preexisting infection at site of needle insertion
* Immunocompromised patients
* Preexisting sensory or motor deficit in operative extremity
* Patient on chronic opioid treatment.
* Patient having a revision of previous ACL reconstruction.
* Pregnancy and lactating women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sobey, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulroy MF, Larkin KL, Batra MS, Hodgson PS, Owens BD. Femoral nerve block with 0.25% or 0.5% bupivacaine improves postoperative analgesia following outpatient arthroscopic anterior cruciate ligament repair. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):24-9. doi: 10.1053/rapm.2001.20773. PMID 11172507
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Mizner RL, Petterson SC, Snyder-Mackler L. Quadriceps strength and the time course of functional recovery after total knee arthroplasty. J Orthop Sports Phys Ther. 2005 Jul;35(7):424-36. doi: 10.2519/jospt.2005.35.7.424. PMID 16108583
- [Background] Johnson RL, Kopp SL, Hebl JR, Erwin PJ, Mantilla CB. Falls and major orthopaedic surgery with peripheral nerve blockade: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):518-28. doi: 10.1093/bja/aet013. Epub 2013 Feb 24. PMID 23440367
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Mudumbai SC, Kim TE, Howard SK, Workman JJ, Giori N, Woolson S, Ganaway T, King R, Mariano ER. Continuous adductor canal blocks are superior to continuous femoral nerve blocks in promoting early ambulation after TKA. Clin Orthop Relat Res. 2014 May;472(5):1377-83. doi: 10.1007/s11999-013-3197-y. PMID 23897505
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Espelund M, Fomsgaard JS, Haraszuk J, Dahl JB, Mathiesen O. The efficacy of adductor canal blockade after minor arthroscopic knee surgery--a randomised controlled trial. Acta Anaesthesiol Scand. 2014 Mar;58(3):273-80. doi: 10.1111/aas.12224. Epub 2013 Nov 8. PMID 24205802
- [Background] Espelund M, Grevstad U, Jaeger P, Holmich P, Kjeldsen L, Mathiesen O, Dahl JB. Adductor canal blockade for moderate to severe pain after arthroscopic knee surgery: a randomized controlled trial. Acta Anaesthesiol Scand. 2014 Nov;58(10):1220-7. doi: 10.1111/aas.12407. PMID 25307707
- [Background] Espelund M, Fomsgaard JS, Haraszuk J, Mathiesen O, Dahl JB. Analgesic efficacy of ultrasound-guided adductor canal blockade after arthroscopic anterior cruciate ligament reconstruction: a randomised controlled trial. Eur J Anaesthesiol. 2013 Jul;30(7):422-8. doi: 10.1097/EJA.0b013e328360bdb9. PMID 23549123
- [Background] Chisholm MF, Bang H, Maalouf DB, Marcello D, Lotano MA, Marx RG, Liguori GA, Zayas VM, Gordon MA, Jacobs J, YaDeau JT. Postoperative Analgesia with Saphenous Block Appears Equivalent to Femoral Nerve Block in ACL Reconstruction. HSS J. 2014 Oct;10(3):245-51. doi: 10.1007/s11420-014-9392-x. Epub 2014 Jun 7. PMID 25264441
- [Background] Andersen HL, Andersen SL, Tranum-Jensen J. The spread of injectate during saphenous nerve block at the adductor canal: a cadaver study. Acta Anaesthesiol Scand. 2015 Feb;59(2):238-45. doi: 10.1111/aas.12451. Epub 2014 Dec 14. PMID 25496028
- [Background] Lewek M, Rudolph K, Axe M, Snyder-Mackler L. The effect of insufficient quadriceps strength on gait after anterior cruciate ligament reconstruction. Clin Biomech (Bristol). 2002 Jan;17(1):56-63. doi: 10.1016/s0268-0033(01)00097-3. PMID 11779647

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants consented but withdrew from the study prior to randomization.
Groups:
- Continuous Adductor Canal Nerve Catheter: Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Patients then undergo general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction with propofol bolus and placement of laryngeal mask airway. Intraoperative opioid limited to no > 150mcg of fentanyl. Completion of procedure, dressing and LMA revoved with patients transferred to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal continuous nerve catheter using normal saline bolus followed by 1/8% bupivacaine infusion through catheter at 8cc/h.
- Long Acting Single Bolus Adductor Canal Nerve Block: Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Patients then undergo general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no > 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine and 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc.
Period: Overall Study
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long Acting Single Bolus Adductor Canal Nerve Block
Started | 34 | 23
Completed | 32 | 21
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Continuous Adductor Canal Nerve Catheter: Ultrasound guided femoral nerve block with 20cc 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal continuous nerve catheter using normal saline bolus followed by 1/8% bupivacaine infusion through catheter at 8cc/h.
  Mepivacaine: 20cc of 2% mepivacaine <20 minutes prior to in room time.
  adductor canal continuous nerve catheter: Placement of ultrasound guided adductor canal continuous nerve catheter
  Normal Saline as bolus followed by bupivacaine: normal
- Long Acting Single Bolus Adductor Canal Nerve Block: Ultrasound guided femoral nerve block with 20cc 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine and 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve.
  Mepivacaine: 20cc of 2% mepivacaine <20 minutes prior to in room time.
  adductor canal nerve block: ultrasound guided adductor canal nerve block
  ropivacaine and dexamethasone: 10cc of 0.5% ropiv
- Total: Total of all reporting groups
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long Acting Single Bolus Adductor Canal Nerve Block | Total
Number analyzed (Participants) | 32 | 21 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 9 | 21
  Between 18 and 65 years | 20 | 12 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 18 | 16 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 21 | 53

OUTCOME MEASURES:

1. Primary Outcome: Subjective Postoperative Pain Scores After Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to Preoperative Femoral Nerve Block Plus Postop Saphenous Nerve Block at 48 Hours After Discharge From PACU.
Description: Subjective subjective postoperative pain scores at POD 2 of preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to preoperative femoral nerve block plus postoperative saphenous nerve block at 48 hours after discharge from PACU using Subjective Numeric Pain Scale score (on an 11 point scale when 0 is no pain and 10 is worst pain).
Time Frame: Post Operative Day 2
Population: Data was unavailable for 1 participant in the Long Acting Single Bolus Adductor Canal Nerve Block group.
Measure: Count of Participants; unit: Participants
Groups:
- Continuous Adductor Canal Nerve Catheter: Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal continuous nerve catheter using normal saline bolus followed by 1/8% bupivacaine infusion through catheter at 8cc/h.
  Mepivacaine: 20cc of 2% mepivacaine <20 minutes prior to in room time.
  adductor canal continuous nerve catheter: Placement of ultrasound guided adductor canal continuous nerve catheter
  Normal Saline as bolus followed by bupivacaine: normal
- Long- Acting Single Bolus Adductor Canal Nerve Block: Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine and 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve.
  Mepivacaine: 20cc of 2% mepivacaine <20 minutes prior to in room time.
  adductor canal nerve block: ultrasound guided adductor canal nerve block
  ropivacaine and dexamethasone: 10cc of 0.5% ropiv
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long- Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 20
Participants
  0 (Pain on Subjective Numeric Pain Scale) | 1 | 1
  1 (Pain on Subjective Numeric Pain Scale) | 2 | 0
  2 (Pain on Subjective Numeric Pain Scale) | 6 | 3
  3 (Pain on Subjective Numeric Pain Scale) | 7 | 4
  4 (Pain on Subjective Numeric Pain Scale) | 5 | 4
  5 (Pain on Subjective Numeric Pain Scale) | 5 | 1
  6 (Pain on Subjective Numeric Pain Scale) | 3 | 2
  7 (Pain on Subjective Numeric Pain Scale) | 2 | 2
  8 (Pain on Subjective Numeric Pain Scale) | 0 | 3
  9 (Pain on Subjective Numeric Pain Scale) | 1 | 0

2. Primary Outcome: Quadriceps Strength of on POD 1 of Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block at 48 Hours After Discharge From PACU
Description: Quadriceps strength on POD 1 of preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to preoperative femoral nerve block plus postoperative saphenous nerve block using Straight Leg Raise Tests, 0-5/5 scale, and knee extension, 0-5/5 scale. On both scales (straight leg raise test and knee extension) 0 indicates the minimum value (low muscle contraction/no movement) and 5 indicates the maximum (normal muscle contraction /pt holds position against pressure).
Time Frame: Post Operative Day 1
Population: Data was unavailable for 1 participant in both groups.
Measure: Count of Participants; unit: Participants
Groups:
- Long-Acting Single Bolus Adductor Canal Nerve Block: Ultrasound guided femoral nerve block with 20cc of 2% mepivacaine <20 minutes prior to in room time. Intraoperative patients will undergo initiation of general anesthesia under the care of the attending anesthesiologist assigned to the patient. Induction will include a propofol bolus and placement of laryngeal mask airway. Intraoperative opioid should be limited to no more than 150mcg of fentanyl. Upon completion of wound closure, appropriate dressing placement, emergence from anesthesia and removal of LMA, patients to be taken to PACU. Once adequately awake and alert this group will receive ultrasound guided adductor canal nerve block with 10cc of 0.5% ropivacaine and 2 mg dexamethasone (0. 5cc), keeping total injectate at 10.5cc to spare significant proximal spread to femoral nerve.
  Mepivacaine: 20cc of 2% mepivacaine <20 minutes prior to in room time.
  adductor canal nerve block: ultrasound guided adductor canal nerve block
  ropivacaine and dexamethasone: 10cc of 0.5% ropiv
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  Straight Leg Raise Test: 0 | 1 | 2
  Straight Leg Raise Test: 1 | 3 | 7
  Straight Leg Raise Test: 2 | 9 | 4
  Straight Leg Raise Test: 3 | 8 | 2
  Straight Leg Raise Test: 4 | 8 | 4
  Straight Leg Raise Test: 5 | 2 | 1
  Knee extension Test: 0 | 2 | 2
  Knee extension Test: 1 | 2 | 3
  Knee extension Test: 2 | 11 | 9
  Knee extension Test: 3 | 9 | 3
  Knee extension Test: 4 | 6 | 2
  Knee extension Test: 5 | 1 | 1

3. Secondary Outcome: Subjective Pain Scores on POD 1 of Patients Receiving (1) Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to (2) Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block
Description: Subjective pain scores on POD 1 of patients receiving (1) preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to (2) preoperative femoral nerve block plus postoperative saphenous nerve block using Subjective Numeric Pain Scale score (on an 11 point scale when 0 is no pain and 10 is worst pain).
Time Frame: Post Operative Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 21
Participants
  0 (Pain on Subjective Numeric Pain Scale) | 1 | 0
  1 (Pain on Subjective Numeric Pain Scale) | 2 | 1
  2 (Pain on Subjective Numeric Pain Scale) | 3 | 1
  3 (Pain on Subjective Numeric Pain Scale) | 11 | 5
  4 (Pain on Subjective Numeric Pain Scale) | 3 | 2
  5 (Pain on Subjective Numeric Pain Scale) | 5 | 2
  6 (Pain on Subjective Numeric Pain Scale) | 4 | 4
  7 (Pain on Subjective Numeric Pain Scale) | 2 | 1
  7.5 (Pain on Subjective Numeric Pain Scale) | 0 | 1
  8 (Pain on Subjective Numeric Pain Scale) | 1 | 4

4. Secondary Outcome: Total Postop Opioid Consumption of Patients Receiving (1) Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to (2) Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block.
Description: Total postop opioid consumption measured by total pain pills on POD 2 and 3 of patients receiving (1) preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to (2) preoperative femoral nerve block plus postoperative saphenous nerve block.
Time Frame: Post Operative Day 2 and 3
Population: Data was unavailable for 1 participant in the Long Acting Single Bolus Adductor Canal Nerve Block group on post operative days 2 and 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 20
Participants
  Post Operative Day 2: 0 pills | 3 | 0
  Post Operative Day 2: 1 pill | 0 | 1
  Post Operative Day 2: 2 pills | 2 | 1
  Post Operative Day 2: 3 pills | 1 | 2
  Post Operative Day 2: 4 pills | 6 | 3
  Post Operative Day 2: 4.5 pills | 0 | 0
  Post Operative Day 2: 5 pills | 9 | 1
  Post Operative Day 2: 6 pills | 2 | 5
  Post Operative Day 2: 7 pills | 2 | 0
  Post Operative Day 2: 8 pills | 6 | 1
  Post Operative Day 2: 9 pills | 0 | 1
  Post Operative Day 2: 10 pills | 1 | 1
  Post Operative Day 2: 11 pills | 0 | 2
  Post Operative Day 2: 12 pills | 0 | 2
  Post Operative Day 2: 13 pills | 0 | 0
  Post Operative Day 3: 0 pills | 3 | 1
  Post Operative Day 3: 1 pill | 1 | 0
  Post Operative Day 3: 2 pills | 3 | 2
  Post Operative Day 3: 3 pills | 3 | 1
  Post Operative Day 3: 4 pills | 6 | 2
  Post Operative Day 3: 4.5 pills | 0 | 1
  Post Operative Day 3: 5 pills | 4 | 4
  Post Operative Day 3: 6 pills | 7 | 2
  Post Operative Day 3: 7 pills | 2 | 0
  Post Operative Day 3: 8 pills | 1 | 2
  Post Operative Day 3: 9 pills | 1 | 0
  Post Operative Day 3: 10 pills | 1 | 1
  Post Operative Day 3: 11 pills | 0 | 1
  Post Operative Day 3: 12 pills | 0 | 2
  Post Operative Day 3: 13 pills | 0 | 1

5. Secondary Outcome: Quadriceps Strength on POD Week 6- Pts Receiving (1) Long-acting Single Bolus Adductor Canal Nerve Block Comparied to (2) Continuous Adductor Canal Nerve Catheter.
Description: Quadriceps strength on POD week 6- pts receiving (1) long-acting single bolus adductor canal nerve block comparied to (2) continuous adductor canal nerve catheter using Straight Leg Raise Tests, 0-5/5 scale, and knee extension, 0-5/5 scale. On both scales (straight leg raise test and knee extension) 0 indicates the minimum value (low muscle contraction/no movement) and 5 indicates the maximum (normal muscle contraction /pt holds position against pressure).
Time Frame: Post Operative Week 6
Population: Data was unavailable for 1 participant in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  Straight Leg Raise Test: 3 | 1 | 1
  Straight Leg Raise Test: 4 | 15 | 9
  Straight Leg Raise Test: 5 | 15 | 10
  Knee extension Test: 3 | 3 | 3
  Knee extension Test: 4 | 21 | 12
  Knee extension Test: 5 | 7 | 5

6. Secondary Outcome: Physical Therapy Participation With a Subjective Assessment of Participant Ability to Participate in PT (Full, Partial, None)
Time Frame: Post Operative Day 1
Population: Data was unavailable for 1 participant in both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  Full participation | 27 | 15
  Partial participation | 4 | 4
  No participation | 0 | 1

7. Secondary Outcome: Subjective Postoperative Pain Score at Post Operative Week 6 of Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block
Description: Subjective postoperative pain score at post operative week 6 of preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to preoperative femoral nerve block plus postoperative saphenous nerve block using Subjective Numeric Pain Scale score with and without activity (on an 11 point scale when 0 is no pain and 10 is worst pain).
Time Frame: Post Operative Week 6
Population: Data was unavailable for 1 participant in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  With activity: 0 (Pain on Subjective Numeric Pain Scale) | 8 | 9
  With activity: 1 (Pain on Subjective Numeric Pain Scale) | 5 | 1
  With activity: 2 (Pain on Subjective Numeric Pain Scale) | 10 | 1
  With activity: 3 (Pain on Subjective Numeric Pain Scale) | 3 | 3
  With activity: 4 (Pain on Subjective Numeric Pain Scale) | 3 | 3
  With activity: 5 (Pain on Subjective Numeric Pain Scale) | 2 | 3
  Without activity: 0 (Pain on Subjective Numeric Pain Scale) | 22 | 14
  Without activity: 1 (Pain on Subjective Numeric Pain Scale) | 4 | 4
  Without activity: 2 (Pain on Subjective Numeric Pain Scale) | 2 | 1
  Without activity: 3 (Pain on Subjective Numeric Pain Scale) | 2 | 1
  Without activity: 4 (Pain on Subjective Numeric Pain Scale) | 1 | 0
  Without activity: 5 (Pain on Subjective Numeric Pain Scale) | 0 | 0

8. Secondary Outcome: Evaluation of Ambulation at Post Operative Week 6 Assessing Independently vs Assistance, With or Without Pain
Time Frame: Post Operative Week 6
Population: Data was unavailable for 1 participant in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  Unassisted with pain | 6 | 6
  Unassisted without pain | 18 | 9
  Assisted with pain | 3 | 2
  Assisted without pain | 4 | 3

9. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Postoperative nausea and vomiting score on POD 1 following discharge from PACU
Time Frame: POD 1 following discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 21
Participants
  No post operative nausea and vomiting | 28 | 17
  Yes post operative nausea and vomiting | 4 | 4

10. Secondary Outcome: Subjective Assessment of Experience With Analgesia
Description: Subjective assessment of experience with analgesia at post operative week 6 using rating of below expectations; met expectations; exceeded expectations
Time Frame: Post Operative Week 6
Population: Data was unavailable for 1 participant in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 31 | 20
Participants
  Below expectations | 0 | 2
  Met expectations | 13 | 7
  Exceeded expectations | 18 | 11

11. Secondary Outcome: Subjective Pain Scores on POD 3 of Patients Receiving (1) Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to (2) Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block
Description: Subjective pain scores on POD 3 of patients receiving (1) preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to (2) preoperative femoral nerve block plus postoperative saphenous nerve block using Subjective Numeric Pain Scale score (on an 11 point scale when 0 is no pain and 10 is worst pain).
Time Frame: Post Operative Day 3
Population: Data was unavailable for 1 participant in the Long Acting Single Bolus Adductor Canal Nerve Block group on post operative day 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 20
Participants
  0 (Pain on Subjective Numeric Pain Scale) | 2 | 2
  1 (Pain on Subjective Numeric Pain Scale) | 3 | 1
  2 (Pain on Subjective Numeric Pain Scale) | 8 | 2
  3 (Pain on Subjective Numeric Pain Scale) | 4 | 5
  4 (Pain on Subjective Numeric Pain Scale) | 6 | 1
  5 (Pain on Subjective Numeric Pain Scale) | 5 | 3
  6 (Pain on Subjective Numeric Pain Scale) | 2 | 3
  7 (Pain on Subjective Numeric Pain Scale) | 2 | 1
  8 (Pain on Subjective Numeric Pain Scale) | 0 | 2

12. Secondary Outcome: Total Postop Opioid Consumption of Patients Receiving (1) Preoperative Femoral Nerve Block Plus Postoperative Continuous Adductor Canal Nerve Catheter Compared to (2) Preoperative Femoral Nerve Block Plus Postoperative Saphenous Nerve Block.
Description: Total postop opioid consumption measured by total pain pills on POD 1 of patients receiving (1) preoperative femoral nerve block plus postoperative continuous adductor canal nerve catheter compared to (2) preoperative femoral nerve block plus postoperative saphenous nerve block.
Time Frame: Post Operative Day1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long-Acting Single Bolus Adductor Canal Nerve Block
Number analyzed (Participants) | 32 | 21
Participants
  0 pills | 1 | 0
  1 pill | 1 | 0
  2 pills | 1 | 0
  3 pills | 3 | 2
  4 pills | 3 | 2
  4.5 pills | 0 | 1
  5 pills | 2 | 4
  6 pills | 8 | 6
  7 pills | 2 | 0
  8 pills | 7 | 3
  10 pills | 2 | 1
  12 pills | 2 | 2

ADVERSE EVENTS:
Time Frame: Time of consent to 6 weeks after surgery (6 weeks)
Description: Complaints and symptoms not existing prior to consent
Arm/Group | Continuous Adductor Canal Nerve Catheter | Long Acting Single Bolus Adductor Canal Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/23
Other Adverse Events (participants affected / at risk) | 3/34 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Adductor Canal Nerve Catheter (N=34) | Long Acting Single Bolus Adductor Canal Nerve Block (N=23)
Leaking from insertion site (Surgical and medical procedures) | 2 (2) | 0 (0)
Knee effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Inflamed esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT02584452/Prot_SAP_000.pdf